CLINICAL TRIAL: NCT02992743
Title: A Pilot Study of NY-ESO-1c259T Cells in Subjects With Advanced Myxoid/ Round Cell Liposarcoma
Brief Title: Letetresgene Autoleucel Engineered T Cells in NY-ESO-1 Positive Participants With Advanced Myxoid/ Round Cell Liposarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208469; ADP-0011-007 (Other: Adaptimmune Therapeutics)
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Results first posted 2022-11-28 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Neoplasms
Keywords: Myxoid/ round cell liposarcoma; Letetresgene autoleucel; Immuno-oncology; T Cell Receptor; Leukapheresis; NY-ESO-1; Adoptive TCR T-cell therapy
MeSH Terms: conditions — Neoplasms; Liposarcoma, Myxoid | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- letetresgene autoleucel (GSK3377794) (Experimental): Eligible participants will be leukapheresed to manufacture engineered T-cells. Participants will then receive letetresgene autoleucel (GSK3377794), as a single intravenous (IV) infusion after completing lymphodepleting chemotherapy.
  Interventions: Drug: letetresgene autoleucel (GSK3377794); Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: letetresgene autoleucel (GSK3377794) — Letetresgene autoleucel (GSK3377794) as an IV infusion.
Drug: Cyclophosphamide — Cyclophosphamide will be used as a lymphodepleting chemotherapy.
Drug: Fludarabine — Fludarabine will be used as a lymphodepleting chemotherapy.

SUMMARY:
This trial will evaluate safety and efficacy of Letetresgene autoleucel (GSK3377794) in participants with advanced myxoid/round cell liposarcoma or high-grade myxoid liposarcoma.

DETAILED DESCRIPTION:
New York esophageal antigen-1 (NY-ESO-1) and LAGE-1a antigens are tumor-associated proteins that have been found in several tumor types. Clinical trials using adoptively transferred T-cells directed against NY-ESO-1/LAGE-1a have shown objective responses. Letetresgene autoleucel (GSK3377794) is the first generation of NY-ESO-1 specific T-cell receptor (TCR) engineered T-cells. This protocol investigates Letetresgene autoleucel treatment in Human Leukocyte Antigen (HLA)-A*02+ participants with NY-ESO1+ advanced myxoid/round cell liposarcoma or high-grade myxoid liposarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Participant is greater than equal to (>=)18 years of age at the time of signing the study informed consent.
* Participant has a diagnosis of advanced (metastatic or inoperable) high grade myxoid liposarcoma / myxoid round cell liposarcoma confirmed histologically and by the presence of the reciprocal chromosomal translocation t(12;16) (q13;p11) or t(12; 22) (q13;q12).
* Participant has measurable disease according to RECIST v1.1 criteria.
* Participant must have previously received or be intolerant to anthracycline based therapy for advanced (metastatic or inoperable) disease.
* Participants who received neoadjuvant/adjuvant anthracycline based therapy and progressed within 6 months of completion of therapy will be eligible.
* Participant must be HLA A*02:01, HLA A*02:05 and/or HLA-A*02:06 positive.
* Participant's tumor (either the most recent archival specimen or a fresh biopsy) is positive for NY-ESO-1 expression by a designated central laboratory.
* Participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Participant has a left ventricular ejection fraction >=45%.
* Participant is fit for apheresis and has adequate venous access for the cell collection.
* Participants must satisfy pregnancy and contraceptive requirements per protocol and have adequate organ function per protocol specified values.

Exclusion Criteria:

* Any previous gene therapy using an integrating vector.
* Any previous allogeneic hematopoietic stem cell transplant.
* Participant has history of allergic reactions attributed to compounds of similar chemical or biologic composition to fludarabine, cyclophosphamide or other agents used in the study.
* Participant has history of chronic or recurrent (within the last year prior to screening) severe autoimmune or immune mediated disease requiring steroids or other immunosuppressive treatments.
* Participant has known active brain or leptomeningeal metastases.
* Participant has other prior malignancy that is not in complete remission.
* Participant has uncontrolled intercurrent illness including, but not limited to:
* (i) Ongoing or active infection.
* (ii) Clinically significant cardiac disease
* (iii) Interstitial lung disease (participants with existing pneumonitis as a result of radiation are not excluded, however, participants must not be oxygen dependent).
* Participant has active infection with Human Immunodeficiency Virus (HIV), Hepatitis B virus (HBV), ), Hepatitis C virus (HCV) or human T-lymphotropic virus (HTLV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] D'Angelo SP, Druta M, Van Tine BA, Liebner D, Schuetze SM, Tap WD, Preston J, Goodison S, D'Souza JW, Kapoor GS, Suchindran S, Zajic S, Bhaskar A, Kaczynski H, Kim J, Klohe E, Corigliano E, Eleftheriadou I, Nathenson MJ, Somaiah N. Letetresgene Autoleucel in Advanced/Metastatic Myxoid/Round Cell Liposarcoma. J Clin Oncol. 2025 May 20;43(15):1777-1788. doi: 10.1200/JCO-24-01466. Epub 2025 Jan 21. PMID 39836945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study evaluating the safety and tolerability of autologous T-Cells expressing enhanced T-cell receptors (TCRs) specific for New York esophageal squamous cell carcinoma (NY-ESO)-1 (letetresgene autoleucel, lete-cel, GSK3377794) in Human Leukocyte Antigen (HLA)-A*02:01, HLA-A*02:05 and/or HLA-A*02:06 participants with Advanced Myxoid/ Round Cell Liposarcoma.
Pre-assignment Details: A total of 23 participants were enrolled in this study. Out of 23 participants, 20 participants received NY-ESO-1c259 T cell infusion.
Groups:
- Reduced Lymphodepletion Dose Plus GSK3377794: Eligible participants were leukapheresed to manufacture autologous NY-ESO-1c259 T cell receptors (TCR) bearing T-cells. Participants underwent lymphodepleting chemotherapy; cyclophosphamide 600 milligrams per meter square per day (mg/m^2/day) plus fludarabine 30 mg/m^2/day on day -7 through day -5 followed by a single infusion of GSK3377794 on Day 1.
- Standard Lymphodepletion Dose Plus GSK3377794: Eligible participants were leukapheresed to manufacture autologous NY-ESO-1^c259 TCR bearing T-cells. Participants underwent lymphodepleting chemotherapy consisting of cyclophosphamide 900 mg/m^2/day starting on day -7 through day -5 plus fludarabine 30 mg/m^2/day on day -8 through day -5 followed by a single infusion of GSK3377794 on Day 1.
Period: Overall Study
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Started | 13 | 10
Received T-cell Infusion | 10 | 10
Completed (Participants who received T-cell infusion and were followed up in this study until death, 15 years post infusion or until transfer to the separate long term follow-up study are considered to have completed.) | 9 (5 participants were transferred to separate long term follow-up study 208750 (NCT03391778) and 4 participants died.) | 8 (8 participants were transferred to separate long term follow-up study 208750 (NCT03391778).)
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death-Prior to T-Cell Infusion | 1 | 0
Not completed — Did Not Meet Inclusion/Exclusion | 1 | 0
Not completed — No measurable disease | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Reduced Lymphodepletion Dose Plus GSK3377794: Eligible participants were leukapheresed to manufacture autologous NY-ESO-1c259 T cell receptors (TCR) bearing T-cells. Participants underwent lymphodepleting chemotherapy; cyclophosphamide 600 mg/m^2/day plus fludarabine 30 mg/m^2/day on day -7 through day -5 followed by a single infusion of GSK3377794 on Day 1.
- Total: Total of all reporting groups
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794 | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 50.0 (6.79) | 46.0 (11.61) | 48.3 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1
  Other: More than one race | 1 | 0 | 1
  White | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Investigator Assessment
Description: Overall response rate (ORR) defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) via investigator assessment per RECIST (Response Evaluation Criteria In Solid Tumors Criteria) v1.1 relative to the total number of participants in the analysis population. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). Confidence intervals (CI) were calculated using the exact (Clopper-Pearson) method.
Time Frame: Up to 24 months
Population: Modified Intent-to-Treat (mITT) population, which included all participants who underwent leukapheresis and received GSK3377794.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Percentage of participants | 20 [2.5 to 55.6] | 40 [12.2 to 73.8]

2. Primary Outcome: Best Overall Response (BOR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Investigator Assessment
Description: The Best Overall Response (BOR) with confirmation for a participant is defined as the best confirmed response (Confirmed Complete Response [CR] > Confirmed Partial Response [PR] > Stable Disease [SD] > Progressive Disease [PD] > Not Evaluable [NE]) from first T cell infusion until disease progression or initiation of new anti-cancer therapy, whichever is earlier, as assessed by the investigator per RECIST v1.1 Criteria.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 2 | 4
  Stable Disease (SD) | 8 | 5
  Progressive Disease (PD) | 0 | 1
  Not Evaluable (NE) | 0 | 0

3. Secondary Outcome: Time to Response (TTR) Assessed by Investigator
Description: Time to response was defined as the interval of time between the date of T-cell infusion and the first documented evidence of the confirmed response (PR or CR), in the subset of participants with a confirmed PR or CR as their best confirmed overall response. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm.
Time Frame: Up to 24 months
Population: Modified Intent-to-Treat (mITT) population which included all participants who underwent leukapheresis and received GSK3377794. Only responders by investigator assessment were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 2 | 4
Months | 1.856 [0.920 to 2.793] | 1.938 [1.889 to 2.366]

4. Secondary Outcome: Duration of Response (DOR) Assessed by Investigator
Description: Duration of response was defined as the interval between the initial date of confirmed response (PR/CR) and the date of progressive disease or death among participants with a confirmed response per RECIST 1.1. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters. Kaplan-Meier Median and 95% confidence intervals are presented. Confidence intervals were calculated using the Brookmeyer-Crowley method.
Time Frame: Up to 24 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 2 | 4
Months | 5.31 [1.87 to 8.74] | 7.47 [6.01 to NA] — Statistics that cannot be calculated due to insufficient events are presented as "NA"

5. Secondary Outcome: Progression Free Survival (PFS) Assessed by Investigator
Description: Progression free survival was defined as the interval between the date of T cell infusion and the earliest date of disease progression or death due to any cause. Progressive disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. PFS based on responses assessed by investigator per RECIST v1.1 is presented. Kaplan-Meier Median and 95% confidence intervals are presented. Confidence intervals were calculated using the Brookmeyer-Crowley method.
Time Frame: Up to 24 months
Population: Modified Intent-to-Treat (mITT) population which included all participants who underwent leukapheresis and received GSK3377794.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Months | 5.36 [2.00 to 11.50] | 8.74 [0.89 to NA] — Statistics that cannot be calculated due to insufficient events are presented as "NA"

6. Secondary Outcome: Best Overall Response (BOR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Independent Reviewer Assessment
Description: The Best Overall Response (BOR) with confirmation for a participant is defined as the best confirmed response (Confirmed Complete Response [CR] > Confirmed Partial Response [PR] > Stable Disease [SD] > Progressive Disease [PD] > Not Evaluable [NE]) from first T cell infusion until disease progression or initiation of new anti-cancer therapy, whichever is earlier, as assessed by independent reviewer per RECIST v1.1 criteria.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 2 | 4
  Stable Disease (SD) | 8 | 3
  Progressive Disease (PD) | 0 | 0
  Not Evaluable (NE) | 0 | 3

7. Secondary Outcome: Overall Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Independent Reviewer
Description: Overall response rate (ORR) defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) via independent reviewer assessment per RECIST v1.1 relative to the total number of participants in the analysis population. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). Confidence intervals (CI) were calculated using the exact (Clopper-Pearson) method.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Percentage of participants | 20 [2.5 to 55.6] | 40 [12.2 to 73.8]

8. Secondary Outcome: Time to Response (TTR) Assessed by Independent Reviewer
Description: as for outcome 3
Time Frame: Up to 24 months
Population: Modified Intent-to-Treat (mITT) population which included all participants who underwent leukapheresis and received GSK3377794. Only responders by independent reviewer were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 2 | 4
Months | 2.366 [1.840 to 2.891] | 1.889 [1.413 to 1.938]

9. Secondary Outcome: Duration of Response (DOR) Assessed by Independent Reviewer
Description: Duration of response was defined as the interval between the initial date of confirmed response (PR/CR) and the date of progressive disease or death among participants with a confirmed response per RECIST 1.1. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm. Kaplan-Meier Median and 95% confidence intervals are presented. Confidence intervals were calculated using the Brookmeyer-Crowley method.
Time Frame: Up to 24 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 2 | 4
Months | NA [NA to NA] — Statistics that cannot be calculated due to insufficient events are presented as "NA" | 7.16 [4.57 to NA] — Statistics that cannot be calculated due to insufficient events are presented as "NA"

10. Secondary Outcome: Progression Free Survival (PFS) Assessed by Independent Reviewer
Description: Progression free survival was defined as the interval between the date of T cell infusion and the earliest date of disease progression or death due to any cause. Progressive disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. PFS based on responses assessed by independent reviewer per RECIST v1.1 is presented. Kaplan-Meier Median and 95% confidence intervals are presented. Confidence intervals were calculated using the Brookmeyer-Crowley method.
Time Frame: Up to 24 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Months | 4.67 [2.79 to NA] — Statistics that cannot be calculated due to insufficient events are presented as "NA" | 9.03 [5.32 to NA] — Statistics that cannot be calculated due to insufficient events are presented as "NA"

11. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAE is defined as any untoward medical occurrence that, at any dose can result in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth or is medically significant or requires intervention to prevent one or the outcomes listed above.
Time Frame: Up to 24 months
Population: Intent-to-Treat (ITT) Population, which included all participants who underwent leukapheresis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 13 | 10
Participants
  SAEs | 5 | 7
  Non-SAEs | 13 | 10

12. Secondary Outcome: Number of Participants With Adverse Event of Special Interest (AESI)
Description: An AESI may be of scientific and medical concern related to the treatment, monitored, and rapidly communicated by investigator to sponsor. The AESI included events of Cytokine release syndrome (CRS), Haematopoietic cytopenias (including pancytopenia and aplastic anaemia), Graft versus host disease (GvHD), Immune Effector-Cell Associated Neurotoxicity Syndrome (ICANS), and Guillain-Barre syndrome.
Time Frame: Up to 24 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Participants
  Participants with any AESI | 10 | 10
  Cytokine release syndrome | 6 | 10
  Haematopoietic cytopenias (including pancytopenia and aplastic anaemia) | 10 | 10

13. Secondary Outcome: Number of Participants With Any Grade Increase in Hematology Results at Worst-case Post-baseline
Description: Blood samples were collected for the analysis of following hematology parameters: hemoglobin, lymphocytes, neutrophils, platelets, leukocytes. Laboratory parameters were graded according to National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 4.0, where Grade1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline is the most recent, non-missing value from a central laboratory within 7 days prior to the lymphodepleting chemotherapy. An increase in grade is defined as an increase in CTCAE grade relative to baseline grade. Data of number of participants with any grade increase at worst-case post-baseline (maximum grade increase post-baseline) is presented.
Time Frame: Up to 24 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Participants
  Hemoglobin Anemia | 9 | 10
  Lymphocyte count decreased | 10 | 10
  Neutrophils | 10 | 10
  Platelets | 9 | 10
  Leukocytes | 10 | 10

14. Secondary Outcome: Number of Participants With Any Grade Increase in Clinical Chemistry Results at Worst-case Post-baseline
Description: Blood samples were collected for the analysis clinical chemistry parameters: glucose, albumin, alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, creatinine, potassium, magnesium, sodium, phosphate, calcium. Laboratory parameters were graded according to National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 4.0, where Grade1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline is the most recent, non-missing value from a central laboratory within 7 days prior to the lymphodepleting chemotherapy. An increase in grade is defined as an increase in CTCAE grade relative to baseline grade. Data of number of participants with any grade increase at worst-case post-baseline (maximum grade increase post-baseline) is presented.
Time Frame: Up to 24 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Participants
  Glucose Hyperglycemia | 5 | 8
  Glucose Hypoglycemia | 1 | 4
  Albumin | 9 | 9
  Alkaline Phosphatase | 4 | 6
  ALT | 7 | 7
  AST | 8 | 8
  Bilirubin: number analyzed (Participants) | 9 | 10
  Bilirubin | 3 | 2
  Creatinine | 4 | 2
  Potassium Hyperkalemia | 1 | 1
  Potassium Hypokalemia | 5 | 9
  Magnesium Hypermagnesemia | 5 | 2
  Magnesium Hypomagnesemia | 2 | 6
  Phosphate | 9 | 10
  Sodium Hypernatremia | 2 | 1
  Sodium Hyponatremia | 8 | 9
  Calcium Corrected for Albumin Hypercalcemia | 2 | 1
  Calcium Corrected for Albumin Hypocalcemia | 1 | 7

15. Secondary Outcome: Number of Participants With Replication Competent Lentivirus (RCL)
Description: RCL was monitored using a polymerase chain reaction (PCR)-based assay that detects and measures copies of the gene coding for the vector's envelope protein, namely vesicular stomatitis virus G protein (VSV-G).
Time Frame: Day 1 (pre-infusion), and at Week 12, Week 24, and 1 year post-infusion
Population: Modified Intent-to-Treat (mITT) population which included all participants who underwent leukapheresis and received GSK3377794.. Only those participants with RCL assessed post T-cell infusion were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 8
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With Insertional Oncogenesis
Description: Peripheral blood mononuclear cells (PBMC) samples were collected for monitoring insertional oncogenesis by PCR for gene modified cells in the blood. DNA from participant identified with >1% PBMC at >=1 year post T-cell infusion was sent for integration site analysis. Integration site analysis was used to assess the possibility of insertional oncogenesis. Participants with insertional oncogenesis were participants with any clones representing >20% of the total.
Time Frame: Up to 2 years
Population: Modified Intent-to-Treat (mITT) population which included all participants who underwent leukapheresis and received GSK3377794. Number of participants analyzed comprises participants for whom integration site analysis was conducted.
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

17. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADAs)
Description: Serum samples were collected to analyze for the presence of ADAs using validated immunoassays.
Time Frame: Up to 24 Months
Population: Modified Intent-to-Treat (mITT) population which included all participants who underwent leukapheresis and received GSK3377794. Only those participants with post-baseline ADA results were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 7 | 10
Participants | 0 | 0

18. Secondary Outcome: Maximum Transgene Expansion (Cmax) of GSK3377794
Description: Cmax was defined as peak cell expansion during the interventional phase. Blood samples were collected to measure Cmax.
Time Frame: Day 2 to Day 15
Population: Modified Intent-to-Treat (mITT) population which included all participants who underwent leukapheresis and received GSK3377794. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies per microgram genomic DNA
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Copies per microgram genomic DNA | 66991.71 (127.0) | 108485.91 (53.4)

19. Secondary Outcome: Time to Cmax (Tmax)
Description: Tmax was defined as time to peak cell expansion during the interventional phase. Blood samples were collected to measure Tmax.
Time Frame: Day 2 to Day 15
Population: as for outcome 18
Measure: Median (Full Range); unit: Days
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Days | 2 [2 to 13] | 4 [2 to 15]

20. Secondary Outcome: Area Under the Time Curve From Zero to Time 28 Days AUC(0-28) of GSK3377794
Description: Area under the cell expansion-time curve from first T-cell infusion to Day 28. Blood samples were collected to measure AUC (0-28 days).
Time Frame: Up to 28 days
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*copies per microgram genomic DNA
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 9 | 9
Days*copies per microgram genomic DNA | 727135.6 (223.9) | 1142798.27 (70.7)

21. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters- PR Interval, QRS Duration, QT Interval, QTcB Interval, QTcF Interval and RR Interval
Description: Triplicate 12-Lead ECGs were collected at baseline visit and single ECGs at other timepoints. At each time point during the study ECG was taken using an ECG machine that automatically calculates the heart rate and measured the PR interval, QRS duration, QTcB, QTcF intervals, RR interval and uncorrected QT interval. Baseline is the most recent, non-missing value within 7 days prior to the lymphodepleting chemotherapy. Change from baseline was to be calculated by subtracting post-dose value from baseline value.
Time Frame: Baseline, Day 1, Day 4 and Day 8
Population: Modified Intent-to-Treat (mITT) population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Milliseconds (msec)
  PR Interval, BASELINE | 152.9 (14.59) | 142 (12.72)
  PR Interval, DAY 1: number analyzed (Participants) | 9 | 9
  PR Interval, DAY 1 | -2.3 (8.66) | -2.2 (9.82)
  PR Interval, DAY 4: number analyzed (Participants) | 9 | 8
  PR Interval, DAY 4 | -10.7 (17.18) | -4 (12.96)
  PR Interval, DAY 8: number analyzed (Participants) | 9 | 8
  PR Interval, DAY 8 | -8.1 (14.9) | 1 (9.32)
  QRS Duration, BASELINE | 91.2 (16.53) | 86.1 (15.01)
  QRS Duration, DAY 1: number analyzed (Participants) | 9 | 9
  QRS Duration, DAY 1 | 2.8 (18.87) | 0.9 (6.49)
  QRS Duration, DAY 4: number analyzed (Participants) | 9 | 8
  QRS Duration, DAY 4 | 2.3 (20.43) | 0.8 (5.75)
  QRS Duration, DAY 8: number analyzed (Participants) | 9 | 8
  QRS Duration, DAY 8 | -2.7 (25.75) | -1 (5.86)
  QT Interval, BASELINE | 401.1 (11.71) | 389.3 (33.57)
  QT Interval, DAY 1: number analyzed (Participants) | 9 | 9
  QT Interval, DAY 1 | -6.4 (23.51) | -8.1 (33.74)
  QT Interval, DAY 4: number analyzed (Participants) | 9 | 8
  QT Interval, DAY 4 | -49.4 (38.59) | -72.5 (47.65)
  QT Interval, DAY 8: number analyzed (Participants) | 9 | 8
  QT Interval, DAY 8 | -16.7 (21.63) | -4.4 (43.41)
  QTcB Interval, BASELINE: number analyzed (Participants) | 2 | 3
  QTcB Interval, BASELINE | 427 (4.24) | 423.3 (19.35)
  QTcB Interval, DAY 1: number analyzed (Participants) | 1 | 3
  QTcB Interval, DAY 1 | 28 (NA) — Number of Participants analyzed was 1 only. | 36.3 (34.03)
  QTcB Interval, DAY 4: number analyzed (Participants) | 2 | 2
  QTcB Interval, DAY 4 | 10 (24.04) | 8 (25.46)
  QTcB Interval, DAY 8: number analyzed (Participants) | 1 | 3
  QTcB Interval, DAY 8 | 1 (NA) — Number of Participants analyzed was 1 only. | 47 (50.27)
  QTcF Interval, BASELINE: number analyzed (Participants) | 8 | 7
  QTcF Interval, BASELINE | 429.9 (23.75) | 425.3 (16.18)
  QTcF Interval, DAY 1: number analyzed (Participants) | 8 | 6
  QTcF Interval, DAY 1 | -10.1 (21.06) | 1.3 (17.36)
  QTcF Interval, DAY 4: number analyzed (Participants) | 7 | 6
  QTcF Interval, DAY 4 | -25.3 (36.62) | 3.3 (31.1)
  QTcF Interval, DAY 8: number analyzed (Participants) | 8 | 5
  QTcF Interval, DAY 8 | -7.5 (22.63) | 16.2 (39.96)
  RR Interval, BASELINE | 842.6 (144.62) | 807.6 (166.39)
  RR Interval, DAY 1: number analyzed (Participants) | 8 | 3
  RR Interval, DAY 1 | -15.8 (98.77) | 5.3 (43.1)
  RR Interval, DAY 4: number analyzed (Participants) | 8 | 2
  RR Interval, DAY 4 | -162.5 (179.21) | -188 (11.31)
  RR Interval, DAY 8: number analyzed (Participants) | 8 | 4
  RR Interval, DAY 8 | -71.6 (109.66) | -138.5 (77.72)

22. Secondary Outcome: Change From Baseline in ECG Mean Heart Rate
Description: Single 12-lead ECG was to be obtained at designated time points during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. Baseline is the most recent, non-missing value within 7 days prior to the lymphodepleting chemotherapy. Change from baseline was to be calculated by subtracting post-dose value from baseline value.
Time Frame: Baseline, Day 1 (Pre-dose), Day 4 and Day 8
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/minute)
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
Number analyzed (Participants) | 10 | 10
Beats per minute (beats/minute)
  BASELINE | 73.0 (12.34) | 78.0 (20.06)
  DAY 1: number analyzed (Participants) | 9 | 9
  DAY 1 | 1.6 (10.08) | 4.8 (14.20)
  DAY 4: number analyzed (Participants) | 9 | 8
  DAY 4 | 20.1 (16.34) | 38.9 (21.95)
  DAY 8: number analyzed (Participants) | 9 | 8
  DAY 8 | 5.4 (12.72) | 9.1 (16.37)

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to 30 months.
Description: All cause mortality, SAEs and non-serious adverse events were reported for the Intent-to-Treat (ITT) population, which included all participants who underwent leukapheresis.
Arm/Group | Reduced Lymphodepletion Dose Plus GSK3377794 | Standard Lymphodepletion Dose Plus GSK3377794
All-Cause Mortality (participants affected / at risk) | 5/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 5/13 | 7/10
Other Adverse Events (participants affected / at risk) | 13/13 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Lymphodepletion Dose Plus GSK3377794 (N=13) | Standard Lymphodepletion Dose Plus GSK3377794 (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 3 (3) | 5 (5)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Lymphodepletion Dose Plus GSK3377794 (N=13) | Standard Lymphodepletion Dose Plus GSK3377794 (N=10)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 9 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Euthyroid sick syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Eye oedema (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (3)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 6 (9)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (11) | 8 (11)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (10) | 5 (5)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 4 (5) | 5 (8)
Fatigue (General disorders) | 8 (9) | 7 (9)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (2)
Malaise (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 4 (5)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 8 (9) | 8 (13)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ocular icterus (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 3 (3) | 6 (8)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (6) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (3)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Culture urine positive (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 10 (24) | 7 (19)
Neutrophil count decreased (Investigations) | 7 (11) | 8 (18)
Platelet count decreased (Investigations) | 4 (5) | 7 (8)
Weight decreased (Investigations) | 1 (2) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 7 (11) | 10 (23)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (7) | 8 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursa disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (5) | 2 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 4 (6)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 4 (4) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Phantom limb syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (4)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (3)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (2)
Hypotension (Vascular disorders) | 3 (4) | 3 (3)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (4) | 3 (3)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02992743/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT02992743/SAP_002.pdf